CLINICAL TRIAL: NCT03747029
Title: Serum Calcium to Phosphorous (Ca/P) Ratio in the Diagnosis of Ca-P Metabolism Disorders: a Multicentre Study
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, Vincenzo Rochira, Associate Professor, Azienda Ospedaliero-Universitaria di Modena
Other Study IDs: 352/17
Record Dates: First submitted 2018-11-16; First posted 2018-11-20 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Phosphorus and Calcium Disorders; Parathyroid Diseases; Hyperparathyroidism; Hypoparathyroidism
MeSH Terms: conditions — Parathyroid Diseases; Hyperparathyroidism; Hypoparathyroidism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with hyperparathyroidism: Patients aged between 18-90 years old with primary hyperparathyroidism. No intervention is provided.
  Interventions: Other: No intervention is provided
- Patients with hypoparathyroidism: Patients aged between 18-90 years old with diagnosed hypoparathyroidism. No intervention is provided.
  .
  Interventions: Other: No intervention is provided
- Control group: Patients that underwent biochemical examination by primary care physician or by endocrinologist in order to assess their calcium-phosphorus metabolism state with normal results.
  No intervention is provided.
  Interventions: Other: No intervention is provided

INTERVENTIONS:
Other: No intervention is provided — No intervention is provided

SUMMARY:
Primary hyperparathyroidism (PHPT) and Hypoparathyroidism (HP) are two of the most frequent disorder of Calcium-Phosphorus (Ca-P) metabolism. The Ca/P ratio is an accurate tool to differentiate patients with PHPT from healthy subjects, according to a previous single-centre study. The reliability of this index is based on the fact that serum Ca and P are inversely related together either in healthy subjects or in patients with PHPT and HP.

DETAILED DESCRIPTION:
The aim of this study is to investigate the accuracy and diagnostic value of Ca/P ratio in the diagnosis of primary hyperparathyroidism and hypoparathyroidism. The definition of a valid cut-off of serum Ca/P ratio for patients with these disorders will be of help especially in those patients with apparently normal biochemical profile, but suggestive for primary hyperparathyroidism and hypoparathyroidism.

ELIGIBILITY:
Inclusion Criteria:

* patients with diagnosis of primary hyperparathyroidism
* patients with diagnosis of hypoparathyroidism
* subjects with normal Calcium-Phosphorus metabolism

Exclusion Criteria for both cases and controls will be:

* age younger than 18 or older than 90 years
* severe renal and liver diseases (i.e. glomerular filtration rate (GFR) <30 ml/min)
* hyperparathyroidism secondary to Vitamin D deficiency
* active metabolic bone disease (e.g. Paget's disease of the bone, osteomalacia, rickets, etc)
* any type of cancer
* malnutrition
* severe obesity (BMI > 40 kg/m2)
* a history of gastrointestinal malabsorption
* sarcoidosis
* hypercortisolism
* diabetes insipidus
* hyperthyroidism
* pseudohypoparathyroidism
* familial hypocalciuric hypercalcemia (FHH)
* treatment with steroids, active forms of vitamin D (calcitriol, ergocalciferol, etc), thiazides, phosphate binders, lithium, cinacalcet, bisphosphonates, and denosumab.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Serum Calcium to Phosphorus ratio will be compared among patients with different disorders of calcium-phosphorus metabolism (primary hyperparathyroidism and hypoparathyroidism) and controls.
Sampling Method: Non-Probability Sample
Enrollment: 1038 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Serum Calcium to Phosphorus ratio | Assessed only once at the diagnosis (from January 2005 to January 2018)
  Calculated formula (serum calcium to serum phosphorus ratio)

SECONDARY OUTCOMES:
Serum Calcium | Assessed only once at the diagnosis (from January 2005 to January 2018)
  From blood sample - Unit of measurement: mg/dl
Serum Phosphorus | Assessed only once at the diagnosis (from January 2005 to January 2018)
  From blood sample - Unit of measurement: mg/dl
Serum Parathormone | Assessed only once at the diagnosis (from January 2005 to January 2018)
  From blood sample - Unit of measurement: pg/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero - Universitaria di Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Madeo B, De Vincentis S, Repaci A, Altieri P, Vicennati V, Kara E, Vescini F, Amadori P, Balestrieri A, Pagotto U, Simoni M, Rochira V. The calcium-to-phosphorous (Ca/P) ratio in the diagnosis of primary hyperparathyroidism and hypoparathyroidism: a multicentric study. Endocrine. 2020 Jun;68(3):679-687. doi: 10.1007/s12020-020-02276-7. Epub 2020 Mar 31. PMID 32236819